CLINICAL TRIAL: NCT02478359
Title: Patient-Centered Physical Activity Coaching in COPD: A Pragmatic Trial
Brief Title: Walk On! Physical Activity Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Huong Q2 Nguyen, Research Scientist, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KPSC IRB 12345
Record Dates: First submitted 2015-06-03; First posted 2015-06-23 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): Standard care patients received their routine care from Kaiser Permanente Southern California and had access to all health services in accordance with their health plan
- Physical Activity Coaching (Walk On!) (Experimental): The 12-month Walk On! intervention included a baseline in-person assessment, collaborative monitoring of steps using two types of activity sensors, semi-automated step goal recommendations using an interactive voice response system or web application, ongoing individualized reinforcement from a physical activity coach, and peer/family support.
  Interventions: Behavioral: Physical Activity Coaching (Walk On!)

INTERVENTIONS:
Behavioral: Physical Activity Coaching (Walk On!) — The 12-month Walk On! intervention included a baseline in-person assessment, collaborative monitoring of steps using two types of activity sensors, semi-automated step goal recommendations using an interactive voice response system or web application, ongoing individualized reinforcement from a physical activity coach, and peer/family support.
  Arms: Physical Activity Coaching (Walk On!)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of the death in the US. The personal, social and economic costs of the disease are tremendous, with annual expenditures of nearly $50 billion, mostly from hospitalizations for exacerbations of COPD and associated sequelae. For the vast majority of patients, despite optimal pharmacological therapy, living with COPD is characterized by unrelieved dyspnea, physical inactivity, deconditioning, and an insidious downward spiral of social isolation and depression that has a profound impact on the lives of patients and their caregivers. There is mounting evidence that physical inactivity is significantly associated with more frequent hospitalizations and increased mortality in COPD even after adjusting for disease severity.

While practice guidelines recommend regular physical activity for all patients with COPD, health systems are challenged in operationalizing an effective and sustainable approach to assist patients in being physically active. The investigators propose a pragmatic randomized controlled trial to determine the effectiveness of a 12-month physical activity coaching intervention (Walk On!) compared to standard care for 1,650 COPD patients from a large integrated health care system.

DETAILED DESCRIPTION:
Physical inactivity is significantly associated with more frequent hospitalizations and increased mortality in COPD even after adjusting for disease severity. While practice guidelines recommend regular physical activity for all patients with COPD, health systems are challenged in operationalizing an effective and sustainable approach to assist patients in being physically active.

A pragmatic randomized controlled trial design will be used to determine the effectiveness of a 12-month home and community-based physical activity coaching intervention (Walk On!) compared to standard care for 2,700 COPD patients from a large integrated health care system. Eligible patients with a COPD-related hospitalization, emergency department visit, or observational stay in the previous 12 months will be automatically identified from the electronic medical records (EMR) system and randomized to treatment arms. The Walk On! intervention includes collaborative monitoring of step counts, semi-automated step goal recommendations, individualized reinforcement from a physical activity coach, and peer/family support.

The primary composite outcome includes all-cause hospitalizations, emergency department visits, observational stays, and death in the 12 months following randomization. Secondary outcomes include COPD-related utilization, cardio-metabolic markers, physical activity, symptoms, and health-related quality of life. With the exception of patient reported outcomes, all utilization and clinical variables will be automatically captured from the EMR.

If successful, findings from this multi-stakeholder driven trial of a generalizable and scalable physical activity intervention model, carefully designed with sufficient flexibility, intensity, duration, and support for a large ethnically diverse sample could re-define the standard of care to effectively address physical inactivity in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any COPD-related hospitalization, emergency department visit or observational stay in the previous 12 months are eligible for the study. COPD-related encounters are defined according to the Centers for Medicare and Medicaid Services (CMS) and National Quality Forum (NQF) criteria for the Hospital Readmission Reduction Program. The following principal discharge diagnoses of COPD (ICD-9 codes: 491.21, 491.22, 491.8, 491.9, 492.8, 493.20, 493.21, 493.22, and 496) or respiratory failure (ICD-9 codes: 518.81, 518.82, 518.84, 799.1) with a secondary diagnosis of COPD exacerbation (ICD-9 codes: 491.21, 491.22, 493.21, 493.22) will be used
* Age >40 years
* On at least a bronchodilator or steroid inhaler prior to the encounter or if not on an inhaler, had a previous COPD diagnosis
* Continuous health plan membership in the 12 months prior to the encounter

Exclusion Criteria:

* FEV1/FVC ratio >0.70 at any point in the past year for those with spirometry data
* Discharged to hospice, a skilled nursing facility, long term-care or another acute care hospital during the index admission
* Level of function at admission or discharge during the index admission is bed bound
* Has Alzheimers disease, dementia or metastatic cancer
* Morbidly obese (BMI >40)
* Completed pulmonary rehabilitation in the last 6 months
* Deceased
* Dis-enrolled from the health plan

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2707 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huong Q Nguyen, PhD, RN, Principal Investigator — Research Scientist
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States

REFERENCES:
- [Background] Nguyen HQ, Bailey A, Coleman KJ, Desai S, Fan VS, Gould MK, Maddock L, Miller K, Towner W, Xiang AH, Moy ML. Patient-centered physical activity coaching in COPD (Walk On!): A study protocol for a pragmatic randomized controlled trial. Contemp Clin Trials. 2016 Jan;46:18-29. doi: 10.1016/j.cct.2015.10.010. Epub 2015 Oct 24. PMID 26597414
- [Background] Nguyen HQ, Moy ML, Fan VS, Gould MK, Xiang A, Bailey A, Desai S, Coleman KJ. Applying the pragmatic-explanatory continuum indicator summary to the implementation of a physical activity coaching trial in chronic obstructive pulmonary disease. Nurs Outlook. 2018 Sep;66(5):455-463. doi: 10.1016/j.outlook.2018.05.005. Epub 2018 Jul 12. PMID 30144938
- [Derived] Nguyen HQ, Moy ML, Liu IA, Fan VS, Gould MK, Desai SA, Towner WJ, Yuen G, Lee JS, Park SJ, Xiang AH. Effect of Physical Activity Coaching on Acute Care and Survival Among Patients With Chronic Obstructive Pulmonary Disease: A Pragmatic Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e199657. doi: 10.1001/jamanetworkopen.2019.9657. PMID 31418811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were randomly assigned 1:1 to Walk On! or Standard Care arm at the point of identification of eligibility based on EMR data.
Pre-assignment Details: Patients assigned to the Walk On! arm were all approached to participate in and consent to the intervention activities.
  Only a randomly selected subgroup within Standard Care (n=537) were approached to complete surveys for comparison with the Walk On! group.
Period: Overall Study
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Started | 1349 | 1358
Intention-to-treat Population Month 12 | 1243 (Disenrolled from health plan: 106) | 1293 (Disenrolled from health plan: 65)
Completed | 1243 | 1293
Not Completed | 106 | 65
Not completed — Disenrolled from health plan | 106 | 65

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!) | Total
Number analyzed (Participants) | 1349 | 1358 | 2707
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 300 | 305 | 605
  >=65 years | 1049 | 1053 | 2102
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (10.14) | 72.4 (10.24) | 72.4 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 739 | 716 | 1455
  Male | 610 | 642 | 1252
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 59 | 81 | 140
  Native Hawaiian or Other Pacific Islander | 6 | 13 | 19
  Black or African American | 188 | 187 | 375
  White | 1021 | 989 | 2010
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 67 | 81 | 148
Region of Enrollment [Number; unit: participants]
  United States | 1349 | 1358 | 2707
Smoking Status [Count of Participants; unit: Participants]
  Never | 162 | 169 | 331
  Former | 933 | 935 | 1868
  Current | 243 | 238 | 481
  Unknown | 11 | 16 | 27
Body mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27 (6) | 27.1 (5.9) | 27.1 (5.9)
Pulmonary Rehabilitation (up to past 3 years) [Count of Participants; unit: Participants] | 82 | 87 | 169
Spirometry - FEV1 % Predicted [Mean (Standard Deviation); unit: %] — Population: Baseline values were not available on EMR for all participants.
  %
    number analyzed (Participants) | 996 | 1040 | 2036
    (all) | 60 (21.9) | 62.1 (23.1) | 61.0 (22.5)
Spirometry - FEV1/FVC ratio [Mean (Standard Deviation); unit: Ratio (X100)] — Population: Baseline values were not available on EMR for all participants.
  Ratio (X100)
    number analyzed (Participants) | 996 | 1040 | 2036
    (all) | 54.8 (14.7) | 55.4 (13.9) | 55.1 (14.3)
Charlson Comorbidity Index score [Count of Participants; unit: Participants] — The total score in the CCI is derived by summing the assigned weights of all comorbid conditions presented by the client. Higher scores indicate a more severe condition and consequently, a worse prognosis
  Participants
    Score 0-2 | 506 | 516 | 1022
    Score 3 | 210 | 231 | 441
    Score 4-5 | 348 | 332 | 680
    Score 6+ | 285 | 279 | 564
Comorbidity [Count of Participants; unit: Participants]
  Heart Failture | 398 | 407 | 805
  Pulmonary Hypertension | 70 | 73 | 143
  Diabetes | 456 | 417 | 873
  Depression | 361 | 380 | 741
  Anxiety | 383 | 359 | 742
  Chronic Pain | 273 | 272 | 545
Medication [Count of Participants; unit: Participants]
  Long-lasting beta-agonists (LABA) | 846 | 800 | 1646
  Long-lasting anticholinergic (LAMA) | 702 | 720 | 1422
  Long-term systemic corticosteroids | 131 | 112 | 243
  Oxygen-use | 550 | 509 | 1059
  Inhaled corticosteroids (ICS) | 1094 | 1053 | 2147
  LAMA & ICS | 631 | 613 | 1244
  LABA & ICS | 844 | 797 | 1641
All Cause Acute Care Utilization in the 12-months Prior to Randomization [Count of Participants; unit: Participants]
  Hospitalizations | 735 | 702 | 1437
  Observation stay | 394 | 392 | 786
  Emergency department visits | 1050 | 1039 | 2089
COPD-Related Acute Care Utilization in the 12-months Prior to Randomization [Count of Participants; unit: Participants]
  Hospitalization | 568 | 539 | 1107
  Observation Stays | 243 | 237 | 480
  Emergency department visits | 766 | 765 | 1531
  Outpatient treated COPD exacerbations | 966 | 936 | 1902

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-cause Hospitalizations, Emergency Department (ED) Visits, Observation Stays, and Deaths
Description: Covariates included in the adjusted multivariate models were age, FEV1% predicted, Charlson comorbidity index, oxygen use, hospitalization for COPD in previous 12 months, outpatient treated COPD exacerbation in previous 12 months, length of time since acute care utilization to randomization, use of LABA or ICS, PA level and study site
Time Frame: 12 months following randomization
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Standard Care: Standard care patients received routine care from Kaiser Permanente Southern California and had access to all health services in accordance with their health plan
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1349 | 1358
Participants | 864 | 883
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.33, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.92 to 1.28]

2. Secondary Outcome: Number of Deaths Among Participants
Description: as for outcome 1
Time Frame: 12 months following randomization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1349 | 1358
Participants | 117 | 117
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.88, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.77 to 1.36]

3. Secondary Outcome: Number of Participants With All-cause Hospitalizations
Description: as for outcome 1
Time Frame: 12 months following randomization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1349 | 1358
Participants | 499 | 502
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.53, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.89 to 1.24]

4. Secondary Outcome: Number of Participants With All-cause Emergency Department Visits
Description: as for outcome 1
Time Frame: 12 months following randomization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1349 | 1358
Participants | 694 | 702
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.73, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.88 to 1.20]

5. Secondary Outcome: Number of Participants With All-cause Observation Stays
Description: as for outcome 1
Time Frame: 12 months following randomization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1349 | 1358
Participants | 269 | 295
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.21, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.93 to 1.37]

6. Secondary Outcome: Number of Participants With COPD-Related Hospitalizations, ED Visits, and Observation Stays
Description: as for outcome 1
Time Frame: 12 months following randomization
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1349 | 1358
Participants | 398 | 411
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.26, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.93 to 1.31]

7. Secondary Outcome: Number of Participants With COPD Exacerbation
Description: COPD exacerbations were ascertained via pharmacy records and utilization data. An outpatient COPD exacerbation will be defined as a care touch (clinic visit, phone, or secure message encounter) with a diagnosis of COPD accompanied by a prescription of either an oral steroid or an antibiotic within 2 days
Time Frame: 12 months following randomization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1349 | 1358
Participants | 706 | 689
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.41, t-test, 2 sided

8. Secondary Outcome: COPD Assessment Test, CAT - 12 Months
Description: The reported mean change between the baseline and 12 Months scores for the Chronic Obstructive Pulmonary Disease Assessment Test (CAT). Score range is 0-40. A negative change score indicates fewer symptoms.
Time Frame: 12 months
Population: As treated population who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 171 | 188
score on a scale
  Baseline | 20.5 (8.47) | 18.0 (7.28)
  12 months | 19.9 (8.03) | 17.8 (7.48)
  Change at 12 months from baseline | -0.56 (6.46) | -0.15 (6.22)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.55, Regression, Linear

9. Secondary Outcome: Physical Activity
Description: Patients were categorized as being: completely inactive (0 mins/week), insufficiently active (1-149 mins/week) or active, meeting national physical activity recommendations (>150 mins/week) of moderate to vigorous physical activity.
Time Frame: 12 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1349 | 1358
Participants
  Inactive (0 mins/wk) Baseline | 890 | 911
  Inactive (0 mins/wk) 12 Months | 819 | 808
  Insufficiently Active (1-149 mins/wk) Baseline | 262 | 245
  Insufficiently Active (1-149 mins/wk) 12 Months | 243 | 268
  Active (>=150 mins/wk) Baseline | 160 | 174
  Active (>=150 mins/wk) 12 Months | 171 | 182
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Covariates included in the adjusted multivariate models were age, FEV1% predicted, Charlson comorbidity index, oxygen use, hospitalization for COPD in previous 12 months, outpatient treated COPD exacerbation in previous 12 months, length of time since acute care utilization to randomization, use of LABA or ICS, PA level and study site; Test type: Superiority; p = 0.34, Regression, Logistic — adjusted p values

10. Secondary Outcome: Personal Health Questionnaire, PHQ8 - 12 Months
Description: The reported mean change between the baseline and 12 Months scores. Score range is 0-24. A negative change score indicates less depressive symptoms.
Time Frame: 12 months
Population: As treated population who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 164 | 183
score on a scale
  Baseline | 6.6 (6.00) | 4.9 (4.22)
  12 months | 6.3 (5.40) | 4.8 (4.10)
  Change at 12 months from Baseline | -0.30 (4.66) | -0.06 (3.90)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.60, Regression, Linear

11. Secondary Outcome: General Anxiety Disorder, GAD-7 - 12 Months
Description: The reported mean change between the baseline and 12 Months scores. Score range is 0-21. A negative change score indicates less anxiety.
Time Frame: 12 months
Population: As treated population who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 164 | 184
score on a scale
  Baseline | 5.2 (5.81) | 4.0 (4.05)
  12 months | 4.5 (5.08) | 3.8 (4.25)
  Changes at 12 months from Baseline | -0.63 (4.44) | -0.21 (3.63)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.32, Regression, Linear

12. Secondary Outcome: PROMIS-10 HRQL , Physical Health - 12 Months
Description: The reported mean change between the baseline and 12 Months T-scores. Score range is 16-68. A positive change score reflects better physical functioning.
Time Frame: 12 months
Population: As treated population who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 172 | 189
score on a scale
  Baseline | 39.8 (8.62) | 40.7 (6.95)
  12 months | 40.3 (8.06) | 41.7 (7.18)
  Change at 12 months from Baseline | 0.49 (6.72) | 0.97 (5.99)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.47, Regression, Linear

13. Secondary Outcome: PROMIS-10 HRQL , Mental Health - 12 Months
Description: The reported mean change between the baseline and 12 Months T-scores. Score range is 21-68. A positive change score reflects better mental health.
Time Frame: 12 months
Population: As treated population who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 172 | 189
score on a scale
  Baseline | 45.3 (8.94) | 47.7 (8.80)
  12 months | 46.0 (8.65) | 47.9 (8.04)
  Changes at 12 months from Baseline | 0.69 (7.39) | 0.26 (6.77)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.33, Regression, Linear

14. Secondary Outcome: Diastolic Blood Pressure
Description: Average of all routine clinic blood pressure reading taken between 6 and 12-months post randomization. BP obtained with temperatures of >100F and those obtained in urgent care were excluded.
Time Frame: 12 months following randomization
Population: ITT population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1127 | 1186
mmHg | 70.5 (9.59) | 70.1 (9.63)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.87, Regression, Linear — Adjusted P value

15. Secondary Outcome: Systolic Blood Pressure
Description: as for outcome 14
Time Frame: 12 months following randomization
Population: ITT population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1127 | 1186
mmHg | 130.8 (14.54) | 130.7 (14.19)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.70, Regression, Linear — Adjusted P value

16. Secondary Outcome: HbA1c Levels
Description: HbA1c levels were obtained only from diabetics and on values closest to the 12 months post randomization
Time Frame: 12 months following randomization
Population: ITT population
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin,
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 412 | 383
percentage of glycosylated hemoglobin, | 7.1 (1.45) | 7.2 (1.36)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.35, Regression, Linear; Adjusted P Values

17. Secondary Outcome: LDL Levels
Description: Cholesterol levels were obtained from values closest to the 12 months post randomization
Time Frame: 12 months following randomization
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 593 | 647
mg/dL | 91.0 (36.96) | 86.6 (32.51)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.09, Regression, Linear — Adjusted P Values

18. Secondary Outcome: HDL Levels
Description: Cholesterol levels were obtained from values closest to the 12 months post randomization
Time Frame: 12 months following randomization
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 620 | 671
mg/dL | 54.3 (18.28) | 53.1 (17.60)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.82, Regression, Linear — Adjusted P Values

19. Secondary Outcome: Total Cholesterol Levels
Description: Cholesterol levels were obtained from values closest to the 12 months post randomization
Time Frame: 12 months following randomization
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 621 | 673
mg/dL | 168.8 (44.91) | 162.3 (41.82)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.16, Regression, Linear — Adjusted P values

20. Secondary Outcome: Triglycerides Levels
Description: Cholesterol levels were obtained from values closest to the 12 months post randomization
Time Frame: 12 months post randomization
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 372 | 429
mg/dL | 128.3 (102.36) | 119.0 (65.60)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.86, Regression, Linear — Adjusted P values

21. Secondary Outcome: Body Mass Index
Description: Body mass index measurements were based on values closest to the 12 months post randomization
Time Frame: 12 months following randomization
Population: ITT population
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1281 | 1302
kg/m^2 | 26.9 (5.94) | 27.07 (5.90)
Statistical Analysis 1: Comparison: Standard Care; Test type: Superiority; p = 0.57, t-test, 2 sided

22. Other Pre Specified Outcome: Number of Participants With All-cause Hospitalization, Emergency Department (ED) Visits, Observation Stays and Deaths
Description: As-treated analyses using logistic regression models that included stabilized propensity score inverse probability of treatment weighting (IPTW) to balance baseline characteristics (socio-demographics, health behaviors, disease severity, comorbidities, inhalers/medications, and health care utilization in the prior year) between patients who participated in Walk On! intervention and the SC group. The first 2 months after randomization were excluded because it was expected that it would take approximately 2 months form the date of randomization to start the intervention.
Time Frame: 2 to 12 months following randomization
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1310 | 321
Participants | 781 | 185
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.69, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.82 to 1.35]

23. Other Pre Specified Outcome: Number of Deaths Among Participants
Description: as for outcome 22
Time Frame: 2 to 12 months following randomization
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1310 | 321
Participants | 95 | 13
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.11, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.35 to 1.11]

24. Other Pre Specified Outcome: Number of Participants With All-cause Hospitalizations
Description: as for outcome 22
Time Frame: 2 to 12 months following randomization
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1310 | 321
Participants | 433 | 91
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.21, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.65 to 1.10]

25. Other Pre Specified Outcome: Number of Participants With All-cause Emergency Department Visits
Description: as for outcome 22
Time Frame: 2 to 12 months following randomization
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1310 | 321
Participants | 610 | 144
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.60, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.84 to 1.36]

26. Other Pre Specified Outcome: Number of Participants With All-cause Observation Stays
Description: as for outcome 22
Time Frame: 2 to 12 months following randomization
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1310 | 321
Participants | 230 | 53
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.63, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.66 to 1.28]

27. Other Pre Specified Outcome: Number of Participants With COPD-Related Hospitalizations, ED Visits, and Observation Stays
Description: as for outcome 22
Time Frame: 2 to 12 months randomization
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1310 | 321
Participants | 195 | 48
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Test type: Superiority; p = 0.80, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.68 to 1.35]

28. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: as for outcome 14
Time Frame: 6-12 months following randomization
Population: As-treated Walk On population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1127 | 300
mmHg | 70.5 (9.59) | 69.6 (8.85)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Covariates included in the as-treated adjusted linear regression analyses were age, FEV1%predicted, Charlson comorbidity index, oxygen use, hospitalization for COPD in previous 12 months, outpatient treated COPD exacerbation in previous 12 months, length of time since acute care utilization to randomization, use of LABA or ICS, PA level, and study site; Test type: Superiority; p = 0.06, Regression, Linear — Adjusted P value

29. Other Pre Specified Outcome: Systolic Blood Pressure
Description: as for outcome 14
Time Frame: 6-12 months following randomization
Population: As-treated Walk On population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 1127 | 300
mmHg | 130.8 (14.54) | 128.8 (13.02)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.07, Regression, Linear — Adjusted P value

30. Other Pre Specified Outcome: HbA1c Levels
Description: HbA1c levels were obtained only from diabetics and on values closest to the 12 months post randomization
Time Frame: 12 months
Population: As-treated Walk On population
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 412 | 97
percentage of glycosylated hemoglobin | 7.1 (1.45) | 7.2 (1.40)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Covariates included in the as-treated adjusted linear regression analyses were FEV1%predicted, Charlson comorbidity index, oxygen use, hospitalization for COPD in previous 12 months, outpatient treated COPD exacerbation in previous 12 months, length of time since acute care utilization to randomization, use of LABA or ICS, PA level, and study site; Test type: Superiority; p = 0.67, Regression, Linear — Adjusted P value

31. Other Pre Specified Outcome: LDL Levels
Description: Cholesterol levels were obtained from values closest to the 12 months post randomization
Time Frame: 12 months
Population: As-treated Walk On population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 593 | 174
mg/dL | 91.0 (36.96) | 85.8 (29.92)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.13, Regression, Linear — Adjusted P value

32. Other Pre Specified Outcome: HDL Levels
Description: Cholesterol levels were obtained from values closest to the 12 months post randomization
Time Frame: 12 months
Population: As-treated Walk On population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 620 | 178
mg/dL | 54.3 (18.28) | 52.8 (16.55)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.34, Regression, Linear — Adjusted P value

33. Other Pre Specified Outcome: Total Cholesterol Levels
Description: Cholesterol levels were obtained from values closest to the 12 months post randomization
Time Frame: 12 months
Population: As-treated Walk On population
Measure: Mean (Standard Deviation); unit: md/dL
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 621 | 178
md/dL | 168.8 (44.91) | 161.4 (38.31)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.11, Regression, Linear — Adjusted P value

34. Other Pre Specified Outcome: Triglycerides Levels
Description: Cholesterol levels were obtained from values closest to the 12 months post randomization
Time Frame: 12 months
Population: As-treated Walk On population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
Number analyzed (Participants) | 372 | 114
mg/dL | 128.03 (102.36) | 116.2 (61.36)
Statistical Analysis 1: Comparison: Standard Care vs Physical Activity Coaching (Walk On!); Covariated included in the as-treated adjusted linear regression analyses were age, FEV1%predicted, Charlson comorbidity index, oxygen use, hospitalization for COPD in previous 12 months, outpatient treated COPD exacerbation in previous 12 months, length of time since acute care utilization to randomization, use of LABA or ICS, PA level, and study site; Test type: Superiority; p = 0.83, Regression, Linear — Adjusted P value

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event monitoring focused on passive monitoring via the EMR, components of the primary composite outcome (all cause hospitalizations, observation stays, emergency department visits, and death) for all randomized patients. Only deaths are reported here as anticipated serious adverse events, not related to study procedures. All-cause acute care utilization events were also considered anticipated serious adverse events, not related to study procedures.
Arm/Group | Standard Care | Physical Activity Coaching (Walk On!)
All-Cause Mortality (participants affected / at risk) | 117/1349 | 117/1358
Serious Adverse Events (participants affected / at risk) | 499/1349 | 502/1358
Other Adverse Events (participants affected / at risk) | 963/1349 | 997/1358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=1349) | Physical Activity Coaching (Walk On!) (N=1358)
All-cause hospitalizations (Investigations) | 499 (499) | 502 (502)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=1349) | Physical Activity Coaching (Walk On!) (N=1358)
Observational Stays (Investigations) | 269 (269) | 295 (295)
Emergency Department Visits (Investigations) | 694 (694) | 702 (702)

LIMITATIONS AND CAVEATS:
It is important to note the low uptake/participation in the Walk On! intervention and its effects on the primary, intention to treat analyses, as well, the sub-optimal baseline and follow-up response rates to the patient-reported outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02478359/Prot_SAP_000.pdf